CLINICAL TRIAL: NCT03818009
Title: Effect of General Anesthesia on Early Postoperative Cognitive Dysfunction in Elective Versus Emergency Cesarean Section
Brief Title: Effect of General Anesthesia on Early Postoperative Cognitive Function in Cesarean Section
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Assistant professor, Beni-Suef University
Other Study IDs: Beni-Suef 17
Record Dates: First submitted 2019-01-20; First posted 2019-01-28 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Anesthesia Morbidity; Cesarean Section Complications
Keywords: Cognitive function postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women undergoing elective CS under general anesthesia: Early postoperative assessment of the cognitive function of patients through evaluation document which will be filled by the anesthesiologist.
  Interventions: Other: Assessment document
- women undergoing emergency CS under general anesthesia: Early postoperative assessment of the cognitive function of patients through evaluation document which will be filled by the anesthesiologist.
  Interventions: Other: Assessment document

INTERVENTIONS:
Other: Assessment document — The anesthesiologist will evaluate through his sheet women's cognitive functions.
  Other Names: Anesthesiologist evaluation sheet

SUMMARY:
Cognitive dysfunction is the impairment of the mental process of perception, memory and information processing. The preoperative cognitive state is important, as mild cognitive impairment may be worsened following a cesarean section. Our study will aim to assess the incidence of early cognitive dysfunction after elective and emergent cesarean section under general anesthesia.

DETAILED DESCRIPTION:
Mechanisms that lead to cognitive decline after anesthesia and surgery remain still unclear and mixed. Some studies suggested that an important role is played by the immune response to surgery. The inflammatory response could contribute to the development of postoperative cognitive decline (POCD0 through secretion of cortisol, cytokines, and other inflammatory mediators. Comparing the effects of general and spinal anesthesia on pregnant patients undergoing an elective cesarean section, found no cognitive change after both anesthesias. Our observational comparative study will be carried out at Beni Suef University Hospital. We will compare early cognitive functions undergoing general anesthesia in patients undergoing elective and emergency cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Women in reproductive age period between 25 and 35 years
* Women booked for an elective or emergency cesarean section.

Exclusion Criteria:

* Mental disorder preoperative
* Medical conditions ( as Hypertension or diabetes or cardiac diseases)

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women in reproductive age period between 25 and 35 years booked for an elective or emergency cesarean section.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
postoperative cognitive decline (POCD) | 3 hours postoperative
  New impairment of memory directly post operative which will be assessed by psychometric questionnaire

SECONDARY OUTCOMES:
impaired performance on intellectual tasks | 3 days postoperative
  New impairment of using mind in daily tasks directly post operative which will be assessed through a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Nesreen Abdel Fattah Abdullah Shehata, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rasmussen LS, O'Brien JT, Silverstein JH, Johnson TW, Siersma VD, Canet J, Jolles J, Hanning CD, Kuipers HM, Abildstrom H, Papaioannou A, Raeder J, Yli-Hankala A, Sneyd JR, Munoz L, Moller JT; ISPOCD2 Investigators. Is peri-operative cortisol secretion related to post-operative cognitive dysfunction? Acta Anaesthesiol Scand. 2005 Oct;49(9):1225-31. doi: 10.1111/j.1399-6576.2005.00791.x. PMID 16146456
- [Result] Wan Y, Xu J, Ma D, Zeng Y, Cibelli M, Maze M. Postoperative impairment of cognitive function in rats: a possible role for cytokine-mediated inflammation in the hippocampus. Anesthesiology. 2007 Mar;106(3):436-43. doi: 10.1097/00000542-200703000-00007. PMID 17325501